CLINICAL TRIAL: NCT00484796
Title: Comparison of Trigeminus-evoked Somatosensory Potentials (TRI-SEP) and Medianus-evoked Somatosensory Potentials (MED-SEP) in Patients Undergoing Carotid Surgery
Brief Title: Trigeminus-evoked Somatosensory Potentials in Patients Undergoing Carotid Surgery
Acronym: TRISEP
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: ISRCTN47041942; ISRCTN47041942
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Carotid Surgery
Keywords: Carotid Surgery; Cerebral Ischemia; Cognitive Deficits; Somatosensory-evoked Potentials; Neuromonitoring
MeSH Terms: conditions — Brain Ischemia; Cognition Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients undergoing carotid surgery
  Interventions: Procedure: MED-SEP; Procedure: TRI-SEP; Procedure: neuropsychological tests

INTERVENTIONS:
Procedure: MED-SEP — intraoperative neurophysiological monitoring
Procedure: TRI-SEP — intraoperative neurophysiologic monitoring
Procedure: neuropsychological tests — neurological short- and longterm outcome

SUMMARY:
Hypothesis: Trigeminus-evoked somatosensory potentials (TRI-SEP) may be used as an alternative technique to medianus-evoked somatosensory potentials (MED-SEP) in patients undergoing elective carotid surgery.

DETAILED DESCRIPTION:
For CNS-monitoring somatosensory-evoked responses ba electrical stimulation of the contralateral median nerve are established: A reduction of amplitude and a delay in latency may represent a sensible marker of imminent cerebral ischemia. This study will evaluate a new concept by using trigeminal nerve evoked somatosensory evoked potentials in comparison to the established MED-SEP. Beside the comparison of two methods of neuromonitoring, this study will investigate the neurological long-term outcome (90-day evaluation) with different neuropsychological tests for the detection of cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Agreement with study procedure
* Elective carotid surgery

Exclusion Criteria:

* Inability to take somatosensory potentials
* Inability to respond to neuropsychological tests
* Severe preoperative neurological deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid surgery
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
detection of episodes of cerebral ischemia during carotid surgery | intraoperative, 28 days, and 60 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Principal Investigator — Klinikum St. Georg, Clinics of Anesthesiology, Critical Care and Pain Therapy
Locations (1):
- Klinikum St. Georg, Clinics of Anesthesiology, Critical Care and Pain Therapy, Leipzig, Saxony, Germany